CLINICAL TRIAL: NCT03209505
Title: The Impact of Contact Lens Coefficient of Friction (CoF) on the Development of Lid Wiper Epitheliopathy (LWE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Eric R. Ritchey, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000386
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Lid Wiper Epitheliopathy
Keywords: Lid Wiper Epitheliopahty; Coefficient of Friction

STUDY DESIGN:
Intervention Model Description: Subjects will be fit in a different contact lens brand in each eye. Assignment of the contact lens to each eye will be randomized. One eye will be fit in a contact lens with a low coefficient of friction while the contralateral eye will be fit in a contact lens with a high coefficient of friction.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be masked to the contact lens brand fit in each eye. The subject's Lid Wiper Epitheliopathy will be graded using photographs of the eyelid, where the grader is masked to the lens type in each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Eye 1: Low coefficient of friction (Other): Subjects will be fit in a different contact lens brand in each eye. Assignment of the contact lens to each eye will be randomized. Eye 1 will be fit in a contact lens with a low coefficient of friction, Acuvue Oasys.
  Interventions: Device: Acuvue Oasys
- Eye 2: High coefficient of friction (Other): Subjects will be fit in a different contact lens brand in each eye. Assignment of the contact lens to each eye will be randomized. Eye 2 One eye will be fit in a contact lens with a high coefficient of friction, Air Optix Night & Day Aqua
  Interventions: Device: Air Optix Night & Day Aqua

INTERVENTIONS:
Device: Acuvue Oasys — FDA approved contact lens, fit for daily wear
  Arms: Eye 1: Low coefficient of friction
Device: Air Optix Night & Day Aqua — FDA approved contact lens, fit for daily wear
  Arms: Eye 2: High coefficient of friction

SUMMARY:
This study examines the development of Lid Wiper Epitheliopathy (LWE) in individuals fit with contact lenses having difference coefficients of friction (CoF)

DETAILED DESCRIPTION:
The primary study objectives are to determine the amount of Lid Wiper Epitheliopathy (LWE) induced in subjects after contact lens fitting that do not have LWE at study enrollment. Subjects in the trial will be fit in 2 contact lenses with different coefficients of friction (CoF). One eye will be fit in a contact lens with a low coefficient of friction (Acuvue Oasys®, Johnson & Johnson Vision, Jacksonville FL) while the contralateral eye will be fit in a contact lens with a high CoF (Air Optix® Night & Day® Aqua, Ft. Worth, TX), as reported in the scientific literature. The eye receiving each lens will be assigned randomly. The presence of LWE will be assessed at 2 different time points, approximately 2 hours after contact lens fitting and approximately after 7 days of contact lens wear.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read and understand the study informed consent
2. Must be a minimum of 18 years of age and less than 46 years of age at study enrollment
3. Must be healthy non-soft contact lens wearers (neophytes), or experienced contact lens wearers that have not worn their contact lenses for a minimum of 7 days
4. Have a spherical equivalent refractive error between -0.75 to -6.50DS at the spectacle plane
5. The subject must be able to attend study visits at the prescribed visit times and adhere to the study instructions

Exclusion Criteria:

1. Pregnant and/or lactating females by self-report
2. Presence of current LWE on the upper eyelid (>0.5 in height or width)
3. Has greater than -1.00DC of refractive cylinder
4. Has greater than 1.00D of anisometropia
5. Is aphakic
6. Has clinically significant corneal or conjunctival staining that would prevent contact lens fitting, as assessed with sodium fluorescein dye
7. Has significant ocular surface disease (e.g. Sjögrens Disease, Stevens-Johnson Syndrome, etc.) or significant Dry Eye Syndrome
8. Has clinically significant corneal vascularization or central corneal scaring
9. Has active ocular surface infection (e.g. conjunctivitis)
10. Has a positive history of eyelid surgery or trauma
11. Has a positive history of refractive surgery
12. Takes medications that significantly impact contact lens comfort and/or ocular surface health
13. Has taken part in another contact lens or contact lens solution clinical trial within the last 7 days
14. Is unwilling to have eyes photographed or video recorded

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Ritchey, OD, PhD, Principal Investigator — University of Houston; Rachel Redfern, OD, PhD, Principal Investigator — University of Houston
Locations (1):
- The Ocular Surface Institute, The University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was a contralateral fitting study with one eye receiving the Acuvue Oasys and the contralateral eye receiving the Air Optix Night and Day. Forty eyes of twenty subjects were examined and completed the study
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Eye 1: Low Coefficient of Friction | Eye 2: High Coefficient of Friction
Started | 10; 20 Eyes | 10; 20 Eyes
Completed | 10; 20 Eyes | 10; 20 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Contact Lenses: Forty (40) eyes of twenty subjects were examined. One eye of each subject was assigned either the low coefficient of friction lens and the other eye received the high coefficient of friction lens. Lens/eye assignment occurred per the study randomization schedule.
Arm/Group | Contact Lenses
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.95 (2.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Refractive Error: Right Eye [Mean (Standard Deviation); unit: Diopters] | -2.19 (1.46)
Refractive Error: Left Eye [Mean (Standard Deviation); unit: Diopters] | -1.94 (1.75)

OUTCOME MEASURES:

1. Primary Outcome: Lid Wiper Epitheliopathy
Description: Lid Wiper Staining of the Upper Eyelid. The lid wiper region of the eyelid is the portion of the marginal conjunctival epithelium that moves across the ocular surface or contact lens during blinking. Participants were classified according to their lid wiper epitheliopathy grade for each eye using the following scale: None = 0, Mild = 0.25 - 1.00, Moderate = 1.25 - 2.00, and Severe = 2.25 - 3.00. Grades range from 0 to 3, where higher grades indicate worsening lid wiper epitheliopathy.
Time Frame: One week post contact lens fitting
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Eye 1: Low Coefficient of Friction | Eye 2: High Coefficient of Friction
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 20 | 20
score on a scale | 0.63 [0.00 to 1.44] | 0.25 [0.00 to 1.94]

2. Secondary Outcome: Lid Wiper Epitheliopathy
Description: as for outcome 1
Time Frame: 2 hours post contact lens fitting
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Eye 1: Low Coefficient of Friction | Eye 2: High Coefficient of Friction
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 20 | 20
score on a scale | 0.75 [0.00 to 1.75] | 0.13 [0.00 to 1.44]

ADVERSE EVENTS:
Time Frame: Date was collected over a 1 week period for each subject.
Arm/Group | Eye 1: Low Coefficient of Friction | Eye 2: High Coefficient of Friction
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03209505/Prot_SAP_000.pdf